CLINICAL TRIAL: NCT06046274
Title: A Phase 2 Exploratory, Multicenter, Open-Label Trial to Determine the Safety and Preliminary Clinical Activity of GEN1046 in Combination With Anticancer Agents in Subjects With Advanced Endometrial Cancer
Brief Title: GEN1046 in Combination With Anticancer Agents for the Treatment of Advanced Endometrial Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment challenged by availability of other treatment options
Sponsor: Genmab (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCT1046-05; 2022-502453-33-00 (EU CTIS Number)
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Advanced Endometrial Cancer
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A: pembrolizumab + acasunlimab (Experimental): Pembrolizumab will be administered in combination with acasunlimab as second-line (2L) or third-line (3L) therapy for dMMR/MSI-H in checkpoint inhibitor (CPI) naïve participants.
  Interventions: Biological: Pembrolizumab; Biological: Acasunlimab
- Cohort B: pembrolizumab + acasunlimab (Experimental): Pembrolizumab will be administered in combination with acasunlimab as 2L or 3L therapy for mismatch repair deficient/ microsatellite instability-high (dMMR/MSI-H) participants who had prior exposure to programmed cell death protein/ programmed death ligand 1 (PD-1/PD-L1) inhibitors.
  Interventions: Biological: Pembrolizumab; Biological: Acasunlimab

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab intravenous (IV) infusion
Biological: Acasunlimab — Acasunlimab IV infusion
  Other Names: GEN1046; DuoBody®-PD-L1x4-1BB

SUMMARY:
The goal of this clinical study is to learn about the bispecific antibody, acasunlimab (also known as GEN1046) in combination with the cancer drug pembrolizumab for treatment of participants with incurable endometrial cancer (cancer of the womb). The main questions the study aims to answer are:

* How well acasunlimab in combination with pembrolizumab works against endometrial cancer
* What are the potential side effects participants may experience when they are treated with acasunlimab in combination with pembrolizumab

Participants will receive both acasunlimab and pembrolizumab. All participants will receive active drug; no one will receive placebo. participants will participate in 1 of 2 cohorts. A participant will receive study treatment up to a maximum of 24 months. The study duration (including screening, treatment, and follow-up) for each participant will be about 39 months.

DETAILED DESCRIPTION:
This is an open-label multicenter study in participants with advanced (unresectable and/or metastatic) endometrial cancer to evaluate the safety and clinical activity of acasunlimab (GEN1046) in combination with immunotherapy.

The trial consists of two cohorts:

* Cohort A (cohort closed)
* Cohort B

The study will enroll approximately 80 participants in Cohort A and B (approximately 40 participants in each cohort).

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically confirmed diagnosis of advanced (unresectable, recurrent, and/or metastatic) endometrial carcinoma that is incurable and for which prior standard first-line treatment has failed.
* Prior to Cycle 1 Day 1 (C1D1), documentation of tumor dMMR/MSI-H status must be available based on local testing.
* Must have progressed on or after at least 1 (but no more than 2) prior line(s) of a systemic chemotherapy regimen for unresectable and/or metastatic endometrial cancer of which at least 1 regimen of platinum-based treatment unless participant is ineligible for or intolerant to platinum.
* Cohort A only: Must be treatment naive for CPIs including PD-1 or PD-L1 inhibitors and other immune CPIs (eg, anti-CTLA-4, anti-LAG3, anti-TIGIT).
* Cohort B only: Must have received and progressed on or after prior treatment with a PD-1/PD-L1 inhibitor alone or in combination. Moreover, the participant's duration of CPI containing treatment and best overall response (BOR) is known, and participant has received a minimum of 2 cycles of CPI.

Exclusion Criteria:

* Histological diagnosis of carcinosarcoma, malignant mixed Műllerian tumor, endometrial leiomyosarcoma, or endometrial stromal sarcomas.
* Ongoing or active infection requiring intravenous treatment with anti-infective therapy, or any ongoing systemic inflammatory condition requiring further diagnostic work-up or management during screening.
* Any prior treatment with any type of antitumor vaccine, or autologous cell immunotherapy.
* Radiotherapy within 14 days prior to first dose of acasunlimab. Note: palliative radiotherapy will be allowed for local pain control under certain conditions.
* Treatment with an anticancer agent, including investigational vaccines within 28 days before or 5 times t1/2, whichever is shorter, prior to the planned first dose of trial treatment or is currently enrolled in an interventional trial.
* Prior treatment with live, attenuated vaccines within 30 days prior to initiation of trial treatment.
* Received granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) support within 4 weeks before the planned first dose of trial treatment.
* Cohort A only: Prior exposure to immune CPIs other than anti-PD-1/anti-PD-L1 (eg, anti-CTLA-4, anti-LAG3, anti-TIGIT) or agents directed at costimulatory T-cell receptors (eg, 4-1BB, OX40)
* Cohort B only:

  * Known history of Grade 3 or higher immune-related adverse events (irAEs) that led to treatment discontinuation of a prior immunotherapy treatment
  * Exposure to any of the following prior therapies/treatments within the specified timeframes:
  * Prior exposure to immune CPIs other than anti-PD-1/anti-PD-L1 (eg, anti-CTLA-4, anti-LAG3, anti-TIGIT) or agents directed at costimulatory T-cell receptors (eg, 4-1BB, OX40)
  * PD-1/PD-L1 antibody within 28 days before the planned first dose of trial treatment

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 4 years
  ORR is defined as the percentage of participants with a confirmed response of partial response (PR) or complete response (CR) according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to 4 years
  DOR is defined for responders as the time from initial onset of response to first progression event, defined as radiographic progression or death as per RECIST v1.1.
Time to Response (TTR) | Up to 4 years
  TTR is defined as the time from first infusion of trial treatment to onset of response as per RECIST v1.1.
Disease Control Rate (DCR) | Up to 4 years
  DCR is defined as the proportion of participants with a confirmed response of PR or CR or stable disease (SD) according to RECIST v1.1.
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and as Per Severity | From first dose date up to 90 days after the study treatment
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product as per CTCAE V5.0. TEAE is defined as an AE occurring or worsening between the first dose of study drug and 30 days after the last dose received.

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (29):
- United States (2):
  - Orlando Health Cancer Institute, Orlando, Florida
  - Rudgers Cancer Institute of New Jersey, New Brunswick, New Jersey
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hospital de Charleroi, Charleroi
  - Universitair Ziekenhuis Ghent, Ghent
  - UZ Leuven, Leuven
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Odense Universitetshospital, Odense
- Italy (5):
  - AOU Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - IRCCS Istituto Europeo di Oncologia IEO, Milan
  - Fondazione G. Pascale, Napoli
  - IRCCS Policlinico Universitario Agostino Gemelli, Roma
  - Ospedale Mauriziano Umberto I, Torino
- South Korea (8):
  - Keimyung University Dongsan Medical Center, Daegu
  - National Cancer Center Korea, Goyang-si
  - Pusan National University, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System|Division of Infectious Diseases, Seoul
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - ICO Girona, Girona
  - Clínica Universidad de Navarra, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundacion Jiménez Díaz, Madrid
  - Clínica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No